CLINICAL TRIAL: NCT03230669
Title: Computer-assisted Delivery of Cognitive Behavioral Therapy for Mental Health and Addictions in Canada
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment and data collection issues
Sponsor: University of Prince Edward Island (Other)
Collaborators: Yale University (Other)
Responsible Party: Principal Investigator, Mary Ann MacSwain, Project Coordinator, University of Prince Edward Island
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6006626
Record Dates: First submitted 2017-07-20; First posted 2017-07-26 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Substance Abuse
Keywords: substance abuse; addiction; etherapy
MeSH Terms: conditions — Substance-Related Disorders; Behavior, Addictive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): this arm receives treatment as usual and no intervention.
- CBT4CBT (Experimental): This arm receives treatment as usual and in addition are given access to an online therapy, cbt4cbt. If placed in this group, individuals are asked to use the online therapy for a minimum of 30 minutes each week for the trial duration of 8 weeks.
  Interventions: Other: cbt4cbt

INTERVENTIONS:
Other: cbt4cbt — This arm receives treatment as usual and in addition are given access to an online therapy, cbt4cbt. If placed in this group, individuals are asked to use the online therapy for a minimum of 30 minutes each week for the trial duration of 8 weeks.
  Arms: CBT4CBT

SUMMARY:
Computer-based Training for Cognitive Behavioural Therapy (CBT4CBT) is a new on-line addiction treatment developed by Dr Kathleen Carroll at the Yale School of Medicine in New Haven, Connecticut. CBT4CBT consists of seven one-hour long online sessions that teach key concepts, including dealing with cravings, problem solving, and decision making skills, to help users reduce substance abuse. CBT4CBT has been rigorously tested throughout various communities in the United States with great success and is currently being rolled out throughout the States. The therapeutic approach of CBT4CBT is unique as its efficacy, durability and cost-savings have been proven in several rigorous clinical trials and will be magnified by the fact that the program can be delivered in Canada, allowing for increased and continual improvements in population health. CBT4CBT has been accepted by both patients and addiction treatment personnel alike and has won numerous clinical innovation awards.

A collaboration has now been formed between Dr Carroll and Drs Michelle Patterson and Juergen Krause of the UPEI Centre for Health and Community Research (CHCR) that will bring CBT4CBT to Canada. While CBT4CBT has previously been tested in urban areas, there are many advantages to offering computer-based training to more rural populations (such as PEI). These more remote areas frequently suffer from a lack of services, as well as a lack of continuity with the services currently offered. CBT4CBT may very well provide that needed continuity to Addictions treatment and has also been shown to improve retention.

DETAILED DESCRIPTION:
CBT4CBT will be the first computer-based, cognitive behavioural therapy program for Addictions treatment to be offered in Canada. CBT4CBT has been rigorously tested in urban populations in the United States but this collaboration will be the first pilot trial in First Nation and other rural communities in Canada. Prince Edward Island has a self-proclaimed need for innovative new substance abuse treatments and CBT4CBT may provide the continuity and retention to traditional therapy programs that current available treatment options often lack. This study will allow CBT4CBT to be tested in several Prince Edward Island communities to gage its efficacy and effectiveness. The results and feedback received from the pilot study will allow the program to be adapted for Canadian populations in order to optimize its positive outcomes within Canada.

CBT4CBT has been tested in urban populations in the United States in three rigorous randomized clinical trials with great success. The nature of CBT4CBT suggests it would also be beneficial in rural and remote populations which are common across Canada. Computer based treatments are cost-effective and although their nature necessitates human participants they have minimal risk associated with them. As the first computer based training for Addictions in Canada this research project could have broad implications for treatment in Addictions across our country.

Analysis techniques will be based on those used in previous CBT4CBT trials conducted by our collaborator, Dr Carroll.

The primary substance abuse outcomes (self-reported abstinence) will be assessed throughout the study and through a six month follow-up. Additional outcomes will include use of other services (medical, legal), patient and provider satisfaction, as well as the costs of implementing the program. Each week, the counsellors will deliver a questionnaire (provided by the CHCR) which covers this range of topics to their patient participating in the trial. The data will be analyzed with a focus on feasibility (retention in both conditions, levels of substance abuse, health problems, and cost by condition).

ELIGIBILITY:
Inclusion Criteria:

* In order to create as representative a sample as possible, the inclusion criteria will be fairly broad, including any consenting individual who reports substance abuse in the past thirty days.
* Individuals who are struggling with substance abuse (the definition of 'abuse' is determined by their counselor).
* Individuals who are 18 years of age or older
* Individuals who have used their substance of choice within the past 28 days.

Exclusion Criteria:

* Individuals who are currently suicidal, homicidal, or require immediate hospitalization will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
primary substance use | 6 months
  Substance use of individuals of their primary drug (or drug of choice)

SECONDARY OUTCOMES:
Secondary substance use | 6 months
  Substance use of individuals including all drugs which are not their drug of choice
Healthcare, social and justice interaction | 6 months
  Use of healthcare, social and justice services by the individuals
CBT4CBT feedback | 8 weeks
  Detailed feedback from experimental group individuals on the cbt4cbt program

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Krause, phd, Principal Investigator — University of Prince Edward Island
Locations (1):
- University of Prince Edward Island, Charlottetown, Prince Edward Island, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-07-20): https://cdn.clinicaltrials.gov/large-docs/69/NCT03230669/Prot_SAP_001.pdf
  • Informed Consent Form (2016-08-08): https://cdn.clinicaltrials.gov/large-docs/69/NCT03230669/ICF_000.pdf